CLINICAL TRIAL: NCT04138537
Title: Olfactory Function and Olfactory Bulb Volume in Acromegaly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20/10.11.10.2017
Record Dates: First submitted 2019-10-23; First posted 2019-10-24 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Acromegaly; Olfactory Disorder
Keywords: Acromegaly; Olfaction; Olfactory disorder
MeSH Terms: conditions — Acromegaly; Anosmia

STUDY DESIGN:
Who Masked: Investigator
Masking Description: OB measurements were done in a single-blinded method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acromegaly group (Other): CCCRC test and OB volume results
  Interventions: Other: OB volume; Other: CCCRC test
- Control Group (Other): CCCRC test and OB volume results
  Interventions: Other: OB volume; Other: CCCRC test

INTERVENTIONS:
Other: OB volume — The mean OB volume was calculated in cubic millimeters and compared between the two groups.
Other: CCCRC test — CCCRC test was done for olfactory function assessment and compared between the two groups.

SUMMARY:
A prospective, controlled, single blinded study was planned. 20 patients with Acromegaly (Acromegaly Group) and 20 healthy subjects (Control Group) were planned to include in the study. Connecticut Chemosensory Clinical Research Center (CCCRC) test was applied to evaluate olfactory functions. Olfactory bulb(OB) volumes were measured with a 1.5 T General Electric Signa Excite MRI scanner.

DETAILED DESCRIPTION:
Acromegaly patients were assessed at the Endocrinology Department for their clinical symptoms, and the nasal examination and olfactory evaluation were done at the Department of Otorhinolaryngology. OB volume was evaluated by a single blinded radiologist. Control group patients that had similar demographical characteristics with the Acromegaly Group were recruited in the study.

The CCCRC test is composed of n-butanol odor threshold test and odor identification test. Olfactory tests were scored out of 7 (0: worst, 7: best olfaction) and mean score was calculated as the total CCCRC test score. OB measurements were done individually on the right and left olfactory bulbs and the mean OB volume was calculated in cubic millimeters.

ELIGIBILITY:
Inclusion Criteria:

* Acromegaly diagnosis
* Healthy subjects that had no nasal problems

Exclusion Criteria:

* Previous nasal surgery
* Acute respiratory tract infection
* Nasal polyposis
* Nasal pathologies that causes nasal obstruction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Olfactory bulb (OB) volume | 18 months
  Measurements were done individually on the right and left OB, and the mean OB volume was calculated in cubic millimeters. The mean OB volume was compared between the two groups.
CCCRC test results | 18 months
  Olfactory tests were scored out of 7 (0: worst, 7: best olfaction) and mean score was calculated as the total CCCRC test score.
  The mean score was compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nazan Degirmenci, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Degirmenci N, Bektas H, Senturk E, Ilhan M, Gunaldi A, Yetis EUM, Eren SB. Changes in olfactory function and olfactory bulb after treatment for acromegaly. Eur Arch Otorhinolaryngol. 2021 Jul;278(7):2357-2362. doi: 10.1007/s00405-020-06515-5. Epub 2021 Jan 2. PMID 33386970